CLINICAL TRIAL: NCT06685861
Title: Effectiveness of Digital Cognitive Behavioral Therapy for the Treatment of Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Shantou University Mental Health Center (Unknown); Hebei Provincial Mental Health Center (Unknown)
Responsible Party: Principal Investigator, Weihua Yue, Professor, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-59
Record Dates: First submitted 2024-11-04; First posted 2024-11-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: i-CBT
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-CBT group (Experimental): i-CBT combined with conventional drug treatment
  Interventions: Device: a digital product based on CBT
- control group (No Intervention): conventional drug treatment

INTERVENTIONS:
Device: a digital product based on CBT — The digital cognitive behavioral therapy in this study is conducted based on a self-developed mobile applet. The therapy is developed by psychotherapists, which is conducted for a total of 8 weeks, with weekly sessions including Al-guided course work and homework.
  Arms: i-CBT group

SUMMARY:
The project proposes to develop a digital product based on cognitive behavioral therapy for the assisted treatment of depression. The digital cognitive behavioral therapy in this study is conducted based on a self-developed mobile applet. The therapy is developed by psychotherapists, which is conducted for a total of 8 weeks, with weekly sessions including AI-guided course work and homework. The aim of this study is to evaluate the therapeutic effect of a digital product based on cognitive behavioral therapy for the assisted treatment of depression in patients through a randomised controlled trial, and to explore its genetic imaging mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-45 years (including 18 and 45), no gender restriction;
2. Meets the diagnostic criteria for depressive disorders according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-Ⅴ);
3. Outpatients or inpatients; Hamilton Depression Rating Scale 17-item (HAMD-17) score ≥ 17; Clinical Global Impressions-Severity (CGI-S) score = 4;
4. Maintenance treatment with antidepressants in the class of Selective Serotonin Reuptake Inhibitors (SSRIs) for at least 4 weeks, or no previous treatment with antidepressants, and can be combined with Lorazepam 0.5mg/dose and Zolpidem Tartrate 5-10mg/n during insomnia and anxiety attacks;
5. Written informed consent obtained from the patient.

Exclusion Criteria:

1. Diagnosed with other mental disorders, including schizophrenia, bipolar disorder, alcohol or substance abuse/dependence, eating disorders, etc.;
2. Individuals with intellectual disabilities or who are unable to cooperate for other reasons, or those lacking or having incomplete civil capacity during the onset of illness;
3. Suffering from neurological or organic brain diseases (such as stroke, cerebral hemorrhage, brain tumors, Parkinson's disease, epilepsy, etc.) and a history of severe traumatic brain injury;
4. Currently undergoing systematic psychological therapy;
5. Individuals who had been treated with convulsion-free electroconvulsive therapy within the last month;
6. Pregnant women or individuals with contraindications to MRI examinations;
7. Individuals who don't know how to use or don't have a smartphone;
8. Individuals with severe suicidal tendencies or at risk of harming others.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Rating Scale (HAMD) | Week 4 and 8 of treatment duration
  The outcome is assessed by 17-item Hamilton Depression Rating Scale (HAMD-17) Scale. Total HAMD scores range from 0 to 52, with higher scores indicating more severe depressive symptoms. The change of HAMD from baseline to 8-week (after intervention) was used as the primary outcome.

SECONDARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) | Week 4 and 8 of treatment duration.
  The outcome is assessed by Montgomery-Asberg Depression Rating Scale (MADRS). Total MADRS score ranges from 0 to 60, with higher scores indicating greater severity of depression. The change of MADRS from baseline to 8-week (after intervention) was used.
Response to treatment | Week 4 and 8 of treatment duration
  Reduction rate of Hamilton Depression Scale (HAMD-17) or Montgomery-Asberg Depression Rating Scale (MADRS) score ≥50% was recognized as response to treatment.
Clinical Global Impression-Severity of Illness (CGI-S) | Week 4 and 8 of treatment duration
  The outcome was assessed by the Clinical Global Impression-Severity of Illness (CGI-S) scale. It is rated on a 7-point scale. Higher scores indicate more severe symptoms.
Change from baseline in Hamilton Anxiety Rating Scale (HAMA) | Week 4 and 8 of treatment duration
  The outcome is assessed by 14-item Hamilton Anxiety Scale (HAMA). Total score ranges from 0 to 56, with higher scores indicating greater severity of anxiety. The change of HAMA from baseline to 8-week (after intervention) was used.
Change from baseline in Ruminative Responses Scale (RRS) | Week 4 and 8 of treatment duration
  This outcome is assessed by Ruminative Responses Scale (RRS). Total score ranges from 22 to 88, with higher scores indicating greater severity of rumination. The change of RRS from baseline to 8-week (after intervention) was used.
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) | Week 4 and 8 of treatment duration
  This outcome is assessed by Pittsburgh Sleep Quality Index (PSQI). Total score ranges from 0 to 21, with higher scores indicating greater severity of sleep problems. The change of PSQI from baseline to 8-week (after intervention) was used.
Change from baseline in Connor-Davidson Resilience Scale (CD-RISC) | Week 4 and 8 of treatment duration
  This outcome is assessed by Connor-Davidson Resilience Scale (CD-RISC). Total score ranges from 0 to 100, with higher scores indicating greater resilience. The change of CD-RISC from baseline to 8-week (after intervention) was used.
Change from baseline in Thinc-Integrated Tool(THINC-it) | Week 8 of treatment duration
  Cognitive function was assessed by Thinc-Integrated Tool(THINC-it) using digital device. The change of THINC-it from baseline to 8-week (after intervention) was used.
Mood Disorder Questionnaire (MDQ) | Week 4 and 8 of treatment duration
  This outcome is assessed by Mood Disorder Questionnaire (MDQ), which is used to assess the positive symptom of bipolar. A positive screening for bipolar disorder is determined when there are ≥7 of the 13 screening symptoms present, at least one "yes" response in the second section indicating the co-occurrence of several symptoms, and a severity level of "moderate" or "serious problem" in the third section.
Rating Scale for Side Effects（SERS） | Week 4 and 8 of treatment duration
  This outcome is assessed by Rating Scale for Side Effects (SERS), which assess 13 side-effects. Total score ranges from 13 to 52, with higher scores indicating more side-effects.
Client Satisfaction Questionnaire-3 （CSQ-3) | Week 8 of treatment duration
  User's satisfaction was assessed by Client Satisfaction Questionnaire-3 （CSQ-3). Total score ranges from 3 to 12. with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hostipal, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No